CLINICAL TRIAL: NCT05858528
Title: Determining Risk Factors for the Development of Psoriatic Arthritis (PsA) Amongst People Living With Psoriasis: A Patient-driven On-line Prospective European Observational Cohort
Brief Title: HIPPOCRATES Prospective Observational Study
Acronym: HPOS
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: 325080
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Psoriatic Arthritis; Psoriasis
Keywords: prognosis; prediction
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bio-samples will be collected from a sub-set of consenting study participants who have either developed PsA or selected study participants who have been identified to be at low or high risk of PsA (using predictive models developed in other studies). Patient centric bio-sample collection will be achieved using self-administered fingerprick blood sampling kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: No intervention in this study
  Interventions: Diagnostic Test: PEST screening questionnaire

INTERVENTIONS:
Diagnostic Test: PEST screening questionnaire — PEST questionnaire to screen for PsA performed every 6 months

SUMMARY:
HIPPOCRATES is an Innovative Medicines Initiative (IMI) funded EU Consortium established to address key unmet clinical needs in psoriatic disease. As part of the project, the HIPPOCRATES Prospective Observational Study (HPOS) is a study of patients with psoriasis which will run across Europe. The study will be led by a research team at University of Oxford and supported by a team at University College Dublin. We are aiming to identify people with psoriasis who are at risk of developing psoriatic arthritis. Up to one-third of patients with psoriasis will develop a related arthritis causing inflammation in the joints and tendons. We want to identify which patients will develop arthritis with the long-term and ambitious aim of trying to prevent the development of arthritis before it occurs. We are recruiting/approaching adults with psoriasis and asking study participants to complete questionnaires every 6 months via a dedicated study website. The questionnaires will include a 'screening questionnaire' to try to identify arthritis. If participants are identified by the 'screening questionnaire' as having possible arthritis, they will be advised to seek local medical help. We will follow up with them to see if they are diagnosed with psoriatic arthritis.

Alongside the questionnaire information from participants, we will ask some participants to provide a blood fingerprick sample using an easy to use at home sampling kit. The blood sample will be posted to a central location (University College Dublin) where it will be stored and then studied in the laboratory to look for markers that may predict the onset of arthritis.

As many (most) participants will not develop arthritis, we are also studying the impact of psoriasis on the participants to learn more about how psoriasis affects people's daily lives across Europe.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a chronic immune-mediated inflammatory disease that affects peripheral joints, entheses and axial sites and which complicates skin and/or nail psoriasis in up to 30% of cases[1]. It is estimated that 1-2% of the general population have PsA and so in the EU between 5 to 10 million people have the disease. It is increasingly recognised that PsA is associated with comorbidities, particularly those which promote the development of accelerated atherosclerosis and contribute to cardiovascular morbidity and mortality[2]. While PsA can be classified using a mixture of clinical, laboratory and radiographic features such as in the ClASsification of Psoriatic ARthritis (CASPAR) criteria[3], evidence suggests that the disease develops for several years before sufficient classifiable clinical features emerge. The evolution from psoriasis to the point at which the patient meets the CASPAR criteria for PsA may occur in stages. These stages include: ① patients with skin and/or nail psoriasis only but with risk factors for subsequent development of PsA; ② an immune activation phase when there is evidence of cytokine (e.g. IL-23/IL-17 and/or TNF) over-production at a cellular or tissue level; ③ a stage where there is asymptomatic evidence of synovio-entheseal inflammation on imaging: MRI or ultrasound; ④ a "prodromal stage" where psoriasis patients may have musculoskeletal symptoms such as arthralgia and/or stiffness but without sufficient signs to make a diagnosis of PsA; and ⑤ PsA meeting CASPAR criteria.

There is an important possibility that some of these stages may be reversible. At present, treatment is focused on those patients who receive a PsA diagnosis (stage ⑤ above) and have ongoing inflammatory disease and evidence of radiographic damage. Future treatment intervention needs to focus on earlier stages of disease so as to limit poor long-term outcomes and possibly prevent the development of PsA. Improving our knowledge of the molecular basis of these stages and the transitions between them will enable us to have a deeper understanding of the progression of psoriasis to PsA.

Using a highly cost-effective strategy, this study will recruit a highly cost-effective and patient-driven prospective European observational cohort of 25,000 psoriasis patients to record demographic and clinical features and selectively collect bio-samples (whole blood, 'plasma'). Adults with psoriasis but without a pre-existing diagnosis of PsA will be recruited via clinics, national and international patient support organisations including those under the umbrella of European Federation of Psoriasis Organisations (EUROPSO), and media campaigns.

The cohort will be managed using an ethically approved secure internet-based platform where participants can register using dynamic consent online. The platform already hosts longitudinal capture of patient reported outcomes measures and is implemented across Europe by the rare bone European Reference Network. The platform also allows feedback of study results to participants.

Data collection will be at baseline with updates every 6 months using the online platform. At each follow up timepoint, participants will complete a validated screening questionnaire for PsA and if they screen positive, they will be advised to seek medical review locally. They will also complete participant (patient) reported outcomes studying the burden of psoriasis. All results will be provided as feedback to the participants. At follow up, participants/patients will also be asked to report if they have been diagnosed with PsA and if they have, to confirm this by uploading a scanned copy or photo of their clinic letter with their diagnosis recorded/stated.

Bio-samples will be collected from a sub-set of consenting study participants who have either developed PsA or selected study participants who have been identified to be at low or high risk of PsA (using predictive models developed in other studies). Patient centric bio-sample collection will be achieved using self-administered fingerprick blood sampling kits.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* Self-reported diagnosis of skin psoriasis (any form)
* Participant is willing and able to give informed consent for participation in the study and complete data in one of the HPOS languages

Exclusion Criteria:

• Pre-existing diagnosis of PsA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with psoriasis but no pre-existing diagnosis of PsA.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of PsA | Up to 3 years
  Development of PsA confirmed by upload of clinic letter confirming diagnosis. As this is a pragmatic study, this will be a local rheumatologist and so the expertise of the physician may vary.

SECONDARY OUTCOMES:
Impact of disease in psoriasis | Up to 3 years
  PsA impact of disease (PsAID)
Functional impact of psoriasis | Up to 3 years
  Multi-dimensional health assessment questionnaire (MD-HAQ)
Depression prevalence in psoriasis | Up to 3 years
  Patient health questionnaire (PHQ-9)
Fatigue impact in psoriasis | Up to 3 years
  FACIT-fatigue
Burden of treatment in psoriasis | Up to 3 years
  Treatment Satisfaction Questionnaire for Medication (TSQM)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Available through HIPPOCRATES consortium
Supporting Information: Study Protocol, SAP, ICF, CSR